CLINICAL TRIAL: NCT07179757
Title: Clinical Outcomes and Quality of Life in Patients With Locally Advanced Vulvovaginal Cancers: Ambispective Registration Study.
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Professor, Radiation Oncology, Gynecology Disease Management Group, Tata Memorial Hospital
Other Study IDs: TMH IEC1 3814
Record Dates: First submitted 2025-08-18; First posted 2025-09-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Vulvo-vaginal Cancer
Keywords: Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: n= 80 Retrospective Cohort
- Cohort B: n=120 Prospective Cohort

SUMMARY:
The vaginal cancers are responsible for 2% of gynecological cancer while vulvar cancers account for 4 % of gynecological cancers. HPV 16 and 33 are most prevalent in vaginal cancers and account for more than half of cases HPV related vaginal cancer. However, adeqaute information is not there. Similarly, structured QOL data is not available for India. Therefore, in the proposed study we will like to systematically evaluate the patterns of relapse and disease outcomes in patients with vulvovaginal cancer treated with radiation (+/- chemotherapy). The therapeutic research in vulvo-vaginal cancers has been relatively slow and such structured registration databases can allow analysis of large number of patients to report on acute and late effect of treatment outcomes using CTCAE and QOL (EORTC QLQ C-30 and VU-34) in rare cancers. We hope that we will get help in identifying thrust areas for future research including prospective interventional trials through this study.

DETAILED DESCRIPTION:
This study will be conducted in two parts:

Retrospective (Cohort A; Waiver of consent requested) This cohort will include patients treated between January 1, 2019 - August 31st, 2021 (or till time of approval of the present IRB application) which will be part of MD thesis of Dr. Priyanshu Tripathi. In these patients only clinic- pathological information will be extracted from the EMR. This cohort will contribute towards the primary objective and secondary endpoints 1 and 2 only. Waiver of consent for this cohort will be applied. Also waiver will be requested for use of available tissue blocks in department of pathology for IHC work. QOL assessment will not be done for this cohort.

Prospective registration study (Cohort B; Study specific consent to be obtained) wherein patients undergoing radical chemo- radiation and details about outcome and pattern of relapse will be studied. This cohort will include patients treated after the IEC approval of this study. These patients will be consented for prospective inclusion of their clinical, pathological, treatment, toxicity and quality of life data collection. . It will be MD thesis of next students. Additionally consent will be obtained for immuno- histochemistry work on the available tissue blocks.

From electronic medical records and radiotherapy information system the details of tumour volume, stage, nodal involvement, baseline hemoglobin,albumin and histological subtype will be obtained. Details of external radiation, concurrent chemotherapy, brachytherapy dose and nodal disease will be obtained. Paper and eCRF will be used to capture data for prospective cohort and only eCRF (SPSS version 20.0)entries will be done for retrospective cohort. Follow up information will be obtained for clinical and radiological evaluations and patterns of relapse in reference to baseline stage will be reported.

Treatment related acute and late sequelae will be recorded using CTCAE version 5.0 For Cohort B longitudinal evaluation of QOL will be performed using the English, Hindi and Marathi version of VU-34 (translations completed with EORTC and Pilot testing project submitted separately) Uni-variate and multivariate analysis will be performed to evaluate impact of various prognostic factors for overall outcome.

Baseline paraffin blocks will be obtained and IHV staining will be performed for p16, AKT and PDL-1 pathway and correlated with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. All patients diagnosed with vulvo- vaginal cancer.
2. Patients treated with Radiation+/- chemotherapy+/-surgery from January 1, 2019- December 31, 2023.

Exclusion Criteria:

1. Patients with Metastatic disease at the presentation.
2. Incomplete information on the EMR.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients who have completed radiation treatment for vulvo-vaginal cancer, and who are undergoing radiation treatment for vulvo-vaginal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
To report patterns of relapse in patients with vulvovaginal cancer treated with radiation (+/- chemotherapy) | 5 years
  To Report pattern of relapse in patients measure by Clinical Examination , By taking folllow up and Symptoms Reporting
To report patterns of disease outcome in patients with vulvovaginal cancer treated with radiation (+/- chemotherapy) | 5 Years
  To Report pattern of relapse in patients measure by Clinical Examination , By taking folllow up and Symptoms Reporting

SECONDARY OUTCOMES:
To report outcomes as a function of p16, AKT, PDL-1 expression. | 5 years
  IHC Staining will be performed for p16, AKT, PDL-1 expression
To report on acute and late effect of treatment outcomes using CTCAE. | 5 years
To report on longitudinal QOL using EORTC QLQ C-30 (English, Hindi, Marathi as applicable) | 5 years
To report on longitudinal QOL using EORTC VU-34 (English, Hindi, Marathi as applicable) | 5 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No